CLINICAL TRIAL: NCT02778581
Title: Randomized, Double Blind, Placebo Controlled Prospective Study, to Evaluate the Effect of a Vegetal Oil in the Disease's Natural Evolution in Patients Diagnosed With Cognitive Impairment or Mild to Moderate Alzheimer Disease.
Brief Title: Study to Evaluate the Effect of a Vegetal Oil on Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Team Foods Colombia S.A. (Industry)
Collaborators: Biopolis S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ALZ-OIL.01
Record Dates: First submitted 2016-05-08; First posted 2016-05-20 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-05

CONDITIONS: Cognitive Impairments; Alzheimer Disease
Keywords: Cognitive Impairment, Alzheimer's Disease, Vegetal Oil
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lipidic Blend 1 (Active Comparator): Glass bottle with 45 ml of vegetal mixture oil. 1 bottle per day
  Interventions: Dietary Supplement: Lipidic Blend 1
- Lipidic Blend 2 (Active Comparator): Glass bottle with 45 ml of vegetal mixture oil. 1 bottle per day
  Interventions: Dietary Supplement: Lipidic Blend 2
- Placebo (Placebo Comparator): Glass bottle with 45 ml of Olive oil. 1 bottle per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lipidic Blend 1 — daily intake of the content of one 45 mL bottle containing the product
  Arms: Lipidic Blend 1
Dietary Supplement: Lipidic Blend 2 — daily intake of the content of one 45 mL bottle containing the product
  Arms: Lipidic Blend 2
Dietary Supplement: Placebo — daily intake of the content of one 45 mL bottle containing olive oil
  Arms: Placebo

SUMMARY:
The aim of the study is to evaluate the beneficial effect of a mixture of vegetal oils with a composition related to short, medium and long unsaturated chain fatty acids on patients with a diagnose of cognitive impairment or mild to moderate Alzheimer disease

DETAILED DESCRIPTION:
The cognitive impairment syndrome is defined as a decrease of the intellectual performance with respect to a previous step in time. The Cognitive impairment has to be considered as a functional alteration with a continuous and physiological evolution in which happen a set of different circumstances:

* A increasing and normal reduction, that appears after the age of sixty, also known as Age-associated memory impairment (AAMI)
* A mild cognitive impairment (MCI), with a recent and mild loss of memory, but higher to that expected because of patient's age and educational level.
* A severe pathological decrease of the mental abilities, also known as, depending on its characteristics: Severe cognitive impairment (SCI), senile dementia and Alzheimer's disease (1).

In the next years it is expected that this disease will become one of the main health and aged-related problem in aged people.(2) Nowadays, there are 35,6 million people with any kind of dementia, and it is estimated that every year, 7,7 million of new patients are diagnosed. (3) The amount of people affected will probably duplicate every 20 years, if effective treatments to stop its evolution are not developed. The forecast estimate up to 81,1 million of patients in 2040, which make this disease in a XXI century real epidemic.(4)

Before reaching the level of dementia, SCI or Alzheimer's disease, the patient will suffer a progressive mild cognitive impairment. In this level, the disease can be early diagnosed and it would be worth to act on it.

Evidences of the Polyunsaturated oils use on the prevention and/or treatment of cognitive impairment.

Polyunsaturated fatty acids (PUFA) can help to improve the cognitive functions. Neuronal tissues, as the brain, retina and the neurone-covering membranes (myelin) include high levels of PUFA. (5) PUFA's act on the order transmission in the Nervous System. Population studies reported the beneficial effect of fish oil, with a high PUFA concentration, on the memory of patients suffering a mild cognitive impairment. (6) It can be also beneficial for Alzheimer's patients, as they are deficient in PUFA's. A diet rich in PUFA'S can improve the cognitive function on patients con cognitive impairment and Alzheimer's disease. (6-8) Epidemiological studies suggest that oils rich in short chain PUFA, should play a beneficial role stopping the initial progression of Alzheimer's disease.

The previous data confirm the possibility of a beneficial effect of the product to study (a mixture of vegetable oils, rich in triglyceride and lecithins) due to the common characteristic of the product with those PUFA's already marketed.

ELIGIBILITY:
Inclusion Criteria:

* informed consents signed by patients and/or caretaker
* The patient has to fulfil dementia clinical criteria.
* Age between 55 and 85 years old.
* MMSE score between 18 and 26.
* The patient can fulfil all neuropsychologic test, according to investigator.
* The patient has to be always with his/her caretaker during monitorization visits
* The caretaker has to be in regular contact with the patient, knowing his/her situation and participation in the study.
* The caretaker has to check four times per week, at least, the product intake, as well as the routine medication and his/her dietetic habits.
* Both caretaker and patient have to be able to complete the product intake during all the length of the study, according to the main investigator.

Exclusion Criteria:

* Patient and/or caretaker not being able to understand and agree in writing their participation in the study.
* Patient disability to oral intake of products.
* Known allergy to any of the product components (active and placebo)
* Evidence of suffering other neuropsychiatric disturbances apart of dementia as: Parkinson disease, psychotic disturbance, bipolar depression.
* regular intake of alcohol higher than 45 g ethanol/day, during the year before study inclusion.
* Any known concurrent malignant pathology in the moment of study inclusion, or severe metabolic, cardiovascular, renal, hepatic, or gastrointestinal disease that cannot allow the ending of the study according the investigator.
* Any analytical abnormality during the screening, apart from: Creatinine no less than 1.7 mg/dL; low levels of Vitamin B12, and TSH abnormal values.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-04 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Changes in Mini-Mental State Examination (MMSE) score | baseline, 3 month, 6 month, 9 month, 12 month
Changes in Global Clinical Dementia Rating (CDR) score | baseline, 3 month, 6 month, 9 month, 12 month

SECONDARY OUTCOMES:
Changes in systemic oxidative parameters in periferic blood samples (Nitric Oxyde) | baseline, 12 month
Changes in systemic oxidative parameters in periferic blood samples (Malondialdehyde (MDA)) | baseline, 12 month
Changes in beta-amyloid protein concentration | baseline, 12 month
  Changes in mean values on high sensitivity beta-amyloid 1-40 and 1-42 protein and TAU-protein in cerebrospinal fluid on those patients with a new diagnose of mild to moderate cognitive impairment, that require an initial lumbar puncture and a new lumbar puncture to control evolution at the end of teh study.
Changes in TAU-Protein concentration | baseline, 12 month
  Changes in mean values on high sensitivity beta-amyloid 1-40 and 1-42 protein and TAU-protein in cerebrospinal fluid on those patients with a new diagnose of mild to moderate cognitive impairment, that require an initial lumbar puncture and a new lumbar puncture to control evolution at the end of teh study.
Changes in regular treatment for the cognitive impairment | baseline, 3 month, 6 month, 9 month, 12 month
Changes in dietetic habits | baseline, 3 month, 6 month, 9 month, 12 month
Changes in Barthel score | baseline, 3 month, 6 month, 9 month, 12 month
Changes in Morisky-Green score | baseline, 3 month, 6 month, 9 month, 12 month
changes in weight | baseline, 3 month, 6 month, 9 month, 12 month
Number of adverse events | baseline, 3 month, 6 month, 9 month, 12 month
  Number of adverse events related or nonrelated to the study or placebo products.

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Navarro-López, MD, Study Director — Universidad Católica San Antonio de Murcia
Locations (2):
- Spain (2):
  - Hospital Universitario Vinalopó, Elche, Alicante
  - Hospital Universitario de Torrevieja, Torrevieja, Alicante

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kueider AM, Parisi JM, Gross AL, Rebok GW. Computerized cognitive training with older adults: a systematic review. PLoS One. 2012;7(7):e40588. doi: 10.1371/journal.pone.0040588. Epub 2012 Jul 11. PMID 22792378
- [Background] Luck T, Luppa M, Briel S, Riedel-Heller SG. Incidence of mild cognitive impairment: a systematic review. Dement Geriatr Cogn Disord. 2010;29(2):164-75. doi: 10.1159/000272424. Epub 2010 Feb 11. PMID 20150735
- [Background] Coronado M, et al. Los ácidos grasos omega-3 y omega-6: Nutrición, bioquímica y salud. REB 25(3) 2006: 72-79
- [Background] Swanson D, Block R, Mousa SA. Omega-3 fatty acids EPA and DHA: health benefits throughout life. Adv Nutr. 2012 Jan;3(1):1-7. doi: 10.3945/an.111.000893. Epub 2012 Jan 5. PMID 22332096
- [Background] Lee LK, Shahar S, Chin AV, Yusoff NA. Docosahexaenoic acid-concentrated fish oil supplementation in subjects with mild cognitive impairment (MCI): a 12-month randomised, double-blind, placebo-controlled trial. Psychopharmacology (Berl). 2013 Feb;225(3):605-12. doi: 10.1007/s00213-012-2848-0. Epub 2012 Aug 30. PMID 22932777
- [Background] Larrieu S, Letenneur L, Berr C, Dartigues JF, Ritchie K, Alperovitch A, Tavernier B, Barberger-Gateau P. Sociodemographic differences in dietary habits in a population-based sample of elderly subjects: the 3C study. J Nutr Health Aging. 2004;8(6):497-502. PMID 15543423
- [Background] Gillette Guyonnet S, Abellan Van Kan G, Andrieu S, Barberger Gateau P, Berr C, Bonnefoy M, Dartigues JF, de Groot L, Ferry M, Galan P, Hercberg S, Jeandel C, Morris MC, Nourhashemi F, Payette H, Poulain JP, Portet F, Roussel AM, Ritz P, Rolland Y, Vellas B. IANA task force on nutrition and cognitive decline with aging. J Nutr Health Aging. 2007 Mar-Apr;11(2):132-52. PMID 17435956
- [Background] Logan AC. Neurobehavioral aspects of omega-3 fatty acids: possible mechanisms and therapeutic value in major depression. Altern Med Rev. 2003 Nov;8(4):410-25. PMID 14653768
- [Background] Bourre JM. Roles of unsaturated fatty acids (especially omega-3 fatty acids) in the brain at various ages and during ageing. J Nutr Health Aging. 2004;8(3):163-74. PMID 15129302
- See also: World Health Organization. Dementia. Fact sheet 362. Published March 2015 — http://www.who.int/mediacentre/factsheets/fs362/en/
- See also: El deterioro cognitivo leve (DCL) en la edad de oro — http://www.uv.es/aprjuv/quaderns/deterioro.pdf